CLINICAL TRIAL: NCT06154824
Title: Repetitive Applications of Pruritogens and Effects of a Cutaneous-induced Pain Stimulation on Nonhistaminergic Itch Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Assistant Professor, Aalborg University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20210046 1st project
Record Dates: First submitted 2023-11-20; First posted 2023-12-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-01

CONDITIONS: Histamine; Cowhage
MeSH Terms: interventions — Histamine

STUDY DESIGN:
Intervention Model Description: The participants will randomly receive 3 consecutive applications of cowhage and histamine.
Who Masked: Participant
Masking Description: Participant will be blinded about application of pruritogens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1st pruritogen (Experimental): The study takes place over two sessions over a period of 7 days. The duration of the sessions is approx. 4 hours in total. In the 1st session, a squared area of 4x4 cm will be selected at the center of each middle forearm of the subject. The two areas will be randomly treated with one of the following substances: cowhage, histamine, BAM 8-22 or vehicle. Each substance will be applied for 10 minutes, during which the pain/itch following the substance application will be monitored. Twenty minutes after each application, the measurements with FLPI will be conducted. Then the measurements of alloknesis and mechanically evoked itch, will be conducted. This procedure will be repeated three times for each substance; so in total each substance will be applied three times, each application lasting 10 minutes.
  Interventions: Other: Cowhage
- 2nd pruritogen (Experimental): The study takes place over two sessions over a period of 7 days. The duration of the sessions is approx. 4 hours in total. In the 1st session, a squared area of 4x4 cm will be selected at the center of each middle forearm of the subject. The two areas will be randomly treated with one of the following substances: cowhage, histamine, BAM 8-22 or vehicle. Each substance will be applied for 10 minutes, during which the pain/itch following the substance application will be monitored. Twenty minutes after each application, the measurements with FLPI will be conducted. Then the measurements of alloknesis and mechanically evoked itch, will be conducted. This procedure will be repeated three times for each substance; so in total each substance will be applied three times, each application lasting 10 minutes.
  Interventions: Other: Histamine

INTERVENTIONS:
Other: Histamine — Histaminergic itch will be evoked by a 1% histamine solution. A droplet of histamine solution will be placed on the predetermined area on the forearm, and the SPT lancet will be pierced through the histamine with 120 g of pressure for 1-2 seconds
  Arms: 2nd pruritogen
Other: Cowhage — 25 spicules will be inserted in the centre of the predefined skin area on the mandibular area. The spicules will be gently rubbed for 15-20 seconds in circular motion to facilitate epidermal penetration
  Arms: 1st pruritogen

SUMMARY:
In This experiment, the investigators would like to test following hypotheses:

repetitive cutaneous administration of pruritogens will lead to a more robust and longer lasting itch sensation compared with a single application. The aim of this project is to investigate a new itch model based on repetitive administration of three different pruritogens: histamine (histaminergic itch), cowhage, and BAM 8-22 (non-histaminergic itch).

DETAILED DESCRIPTION:
Chronic itch affects approximately a fifth of the global population and is associated with substantial negative consequences for the affected individuals. Furthermore, there is a lack of efficient treatment options for chronic itch. In order to mimic a clinical itch condition as presented in patients, the aim of the project is to investigate a new itch model based on repetitive administration of three different pruritogens: histamine (histaminergic itch), cowhage, and BAM 8-22 (non-histaminergic itch). The hypothesis is that repetitive cutaneous administration of pruritogens will lead to a more robust and longer-lasting itch sensation compared with a single application. This proposal for a new itch model could better mimic clinical itch conditions and be used to investigate fundamental mechanisms, new anti-pruritic drugs, and their possible mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other addictive drugs
* Previous or current history of neurological (e.g. neuropathy), immunological (e.g. asthma, immune deficiencies, arthritis) musculoskeletal (e.g. muscular pain in the upper extremities,), cardiac disorder, or mental illnesses that may affect the results
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamines, antipsychotics, and pain killers, as well as systemic or topical steroids
* Skin diseases (e.g. atopic dermatitis, pruritus nodularis, eczema, psoriasis)
* Moles, scars, or tattoos in the area to be treated or tested.
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within one week of study entry (four weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Assessment of itch intensity | 1 minute post itch provocation
  Immediately following the itch provocations, participants will be instructed to rate the itch intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no itch' and 100 'worst itch imaginable'.
Assessment of pain intensity | 1 minute post itch provocation
  Immediately following the itch provocations, participants will be instructed to rate the pain intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no pain' and 100 'worst pain imaginable'.

SECONDARY OUTCOMES:
Superficial blood perfusion | 10 minutes post itch provocation
  The evoked cutaneous inflammation (quantified by superficial blood perfusion) will be measured by full-field laser perfusion imaging.
Alloknesis | 12 minutes post itch provocation
  Alloknesis sensation is measured using a standardized sensory brush (SENSELab Brush-05, Somedic AB, Hörby, Sweden) exerting a force of 200 to 400 mN.
Mechanically evoked itch | 15 minutes post itch provocation
  Mechanically evoked itch is measured using three von Frey filaments of 4.08, 4.16 and 4.31 (1.0, 1.4, 2.0 g, respectively) (North Coast Medical, Gilroy, CA). The center of the skin area is stimulated by 3 pricks, repeated 3 times in short succession. After a total of 9 stimulations, the participants will report the itch elicited on a numerical rating scale (NRS) from 0 to 10 (0 = "no itch"; 10 = "worst imaginable itch").

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No